CLINICAL TRIAL: NCT04166916
Title: Modulation of Sleep Slow Wave Activity Through Acoustic Stimulation and Its Consequences on Cardiovascular Functions
Brief Title: Role of Sleep in Cardiovascular Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Caroline Lustenberger (Other)
Responsible Party: Sponsor-Investigator, Caroline Lustenberger, Principal Investigator, Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2019-01538
Record Dates: First submitted 2019-10-18; First posted 2019-11-18 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Sleep
MeSH Terms: interventions — Acoustic Stimulation

STUDY DESIGN:
Intervention Model Description: we forecast the enrollment of 70 participants which includes the conduction of pilot assessments and the collection of 18 complete participant datasets for the main clinical trial (described here).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Slow waves enhancing acoustic stimulation (Active Comparator): During non-rapid eye movement (NREM) sleep, acoustic stimuli will be played to increase slow wave amplitude.
  Interventions: Other: Acoustic stimulation
- SHAM: no application of acoustic stimuli (Sham Comparator): During NREM sleep no acoustic stimuli will be played.
  Interventions: Other: SHAM acoustic stimulation
- Slow waves decreasing acoustic stimulation (Active Comparator): During NREM sleep acoustic stimuli will be played to decrease/modulate slow waves amplitude in a dose-dependent way (e.g. less pronounced than arm 1).
  Interventions: Other: Acoustic stimulation

INTERVENTIONS:
Other: Acoustic stimulation — Acoustic stimulation to modulate slow waves.
  Arms: Slow waves decreasing acoustic stimulation; Slow waves enhancing acoustic stimulation
Other: SHAM acoustic stimulation — This is the sham-control intervention; only the biosignal will be recorded but no acoustic stimulation will be played.
  Arms: SHAM: no application of acoustic stimuli

SUMMARY:
Sleep and particularly deep sleep are playing an important role for brain and body health. Poor sleep has been associated with risk factors for cardiovascular disease and moreover, is hypothesized to increased mortality risk of cardiovascular diseases. Yet, the role of specific sleep processes for cardiovascular function remains unclear. Particularly deep sleep, which is manifested by large amplitude, low frequency oscillations is of importance for the restorative functions of sleep. Thus, the modulation of deep sleep by auditory stimulation will be of central interests to assess the cause-effect relationship of specific processes within sleep for cardiovascular regulation.

This study will assess the effects of slow wave modulating auditory stimulation on cardiovasuclar functions in healthy male participants.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* Good general health status
* Male subjects 18-84 years of age
* Native German speaker or good understanding of German

Exclusion Criteria:

* Contraindications on ethical grounds,
* Known or suspected non-compliance, drug or alcohol abuse,
* Regular medication intake that could pronouncedly affect outcomes of interest (e.g. beta-blocker)
* Long (> 9.5 hours per night) or short sleepers (< 6.5 hours per night),
* Smoking (regular smoker, >10 days per year, smoking not allowed during study participation)
* Participation in another study with investigational drug/therapy/interventions within the 30 days preceding and during the present study (start date adapted accordingly),
* Diseases or lesions of the nervous system (acute or residual included neurological and psychiatric diseases),
* Clinically significant concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, etc.),
* Pacemaker,
* Intake of on-label sleep medication,
* Presence or suspicion of sleep disorders (e.g., insomnia, sleep disordered breathing (apnea), restless legs syndrome). Possibility of apnea might be assessed in the screening night,
* Body Mass Index < 18 or > 30 kg/m2,
* Irregular sleep-wake rhythm (e.g. shift working),
* Bad sleep quality during screening night (e.g. < 75% sleep efficiency in screening night)
* Significant sleep complaints in general or excessive daytime sleepiness (PSQI > 5; ESS ≥ 11),
* Travelling more than 2 time zones in the 2 weeks before experimental session starts or during intervention (start of experiment will be adapted to fit with this criteria),
* Hearing disability/ hearing aid (only an exclusion if in a simple audiometry participants cannot hear intervention tone sound levels),
* Skin disorders/problems/allergies (face region) that will significantly worsen with electrode application,
* High caffeine consumption (> 5 servings/day; including coffee and caffeinated energy drinks),

Ages: 18 Years to 84 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2020-01-13 (Actual); Primary Completion 2021-03-11 (Actual); Study Completion 2021-03-11 (Actual)

PRIMARY OUTCOMES:
Cardiac autonomic regulation | continuously across approximately 8 hours of sleep with and without acoustic stimulation
  assessed by heart rate variability derived from electrocardiography
Change in cardiac autonomic regulation | Before to after approximately 8 hours of sleep with and without acoustic stimulation
  assessed by changes in heart rate variability derived from electrocardiography
Heart rate | continuously across approximately 8 hours of sleep with and without acoustic stimulation
  measured with electrocardiography
Change in heart rate | Before to after approximately 8 hours of sleep with and without acoustic stimulation
  measured with electrocardiography
Marker for sleep depth | continuously across approximately 8 hours of sleep with and without acoustic stimulation
  Slow wave activity assessed with high-density electroencephalography(hdEEG)

SECONDARY OUTCOMES:
Change in vascular functioning | Before and/or after approximately 8 hours of sleep with and without acoustic stimulation
  Assessed by outcomes of blood profiles of vascular inflammation, pulmonal arterial pressure, intima media thickness, or echocardiography
Arterial pressure waveform | continuously across approximately 8 hours of sleep with and without acoustic stimulation
  assessed by arterial pressure waveform measures
Change in arterial pressure waveform | Before to after approximately 8 hours of sleep with and without acoustic stimulation
  assessed by arterial pressure waveform measures
Oxyen saturation | continuously across approximately 8 hours of sleep with and without acoustic stimulation
  assessed by pulse oximetry
Overnight memory consolidation | Before to after approximately 8 hours of sleep with and without acoustic stimulation
  Assessed by memory tasks
Changes in vigilance | Before to after approximately 8 hours of sleep with and without acoustic stimulation
  assessed by simple vigilance task
Changes in muscular fatigue | Before to after approximately 8 hours of sleep with and without acoustic stimulation
  assessed by simple muscular fatigue task
Changes in bandwidth of of 0.5-30 Hz of high-density electroencephalography (hdEEG) | Before to after approximately 8 hours of sleep with and without acoustic stimulation
  Assessment of resting state and task-related hdEEG
Hypnogram | Over approximately 8 hours of sleep with and without acoustic stimulation
  assessed by sleep staging of hdEEG data

OTHER OUTCOMES:
Incidence of Intervention-related Adverse Events (Safety and Tolerability) | Through study completion approximately one month
  Any adverse or serious adverse event during the study period will be assessed
Chronotype | During initial screening session before start of experimental period (single-time assessment during one initial 1-day visit)
  Assessment of circadian type
Body mass index | During initial screening session before start of experimental period (single-time assessment during one initial 1-day visit)
  Assessment of height, weight to calculate body mass index
Hip-to-waist ratio | During initial screening session before start of experimental period (single-time assessment during one initial 1-day visit)
  Assessment of hip and waist circumference to calculate hip-to-waist ratio
Subjective sleep quality | During initial screening session before start of experimental period (single-time assessment during one initial 1-day visit)
  assessed by Pittsburgh Sleep quality index
Daytime sleepiness | During initial screening session before start of experimental period (single-time assessment during one initial 1-day visit)
  assessed by Epworth sleepiness scale
Change in sleepiness | Before to after approximately 8 hours of sleep with and without acoustic stimulation
  assessed by Karolinska Sleepiness Scale or Stanford Sleepiness Scale
Body composition | During initial screening session before start of experimental period (single-time assessment during one initial 1-day visit)
  Assessment of body composition through DEXA scan

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Lustenberger, PhD, Principal Investigator — ETH Zurich
Locations (1):
- ETH Zurich, Zurich, Schweiz, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huwiler S, Carro-Dominguez M, Stich FM, Sala R, Aziri F, Trippel A, Ryf T, Markendorf S, Niederseer D, Bohm P, Stoll G, Laubscher L, Thevan J, Spengler CM, Gawinecka J, Osto E, Huber R, Wenderoth N, Schmied C, Lustenberger C. Auditory stimulation of sleep slow waves enhances left ventricular function in humans. Eur Heart J. 2023 Oct 21;44(40):4288-4291. doi: 10.1093/eurheartj/ehad630. No abstract available. PMID 37794725